CLINICAL TRIAL: NCT07267156
Title: Evaluation of a New Postoperative Dressing After Hallux Valgus Surgery
Acronym: psmt3D
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Assal for Foot Medicine and Surgery SA (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 2025-00900
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Hallux Valgus
Keywords: Hallux valgus; Postoperative dressing
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3D-printed spacer (Experimental): 3D-printed spacer
  Interventions: Device: Custom 3D-printed toe spacer
- Standard Folded-Gauze Spacer (Active Comparator): Participants receive a standard postoperative toe spacer consisting of folded medical gauze placed between the hallux and second toe immediately after surgery. The spacer is worn continuously for 5 weeks as part of routine care and represents the current standard method used at the study center.
  Interventions: Device: Standard folded-gauze toe spacer

INTERVENTIONS:
Device: Custom 3D-printed toe spacer — A custom-made spacer designed to maintain hallux alignment after bunion surgery. It is produced individually for each participant using 3D-printing technology based on foot measurements. The device is manufactured from thermoplastic polyurethane (TPU), a biocompatible material commonly used for orthopedic applications. The spacer is externally applied between the hallux and second toe immediately following surgery and remains in place continuously for 5 weeks as part of routine postoperative care. The device does not contact the surgical wound, which is covered by a sterile dressing, and does not require any additional medical procedures for application or removal.
  Arms: 3D-printed spacer
Device: Standard folded-gauze toe spacer — Participants receive a standard postoperative toe spacer consisting of folded medical gauze placed between the hallux and second toe immediately after surgery. The spacer is worn continuously for 5 weeks as part of routine care and represents the current standard method used at the study center.
  Arms: Standard Folded-Gauze Spacer

SUMMARY:
Hallux valgus, commonly known as a bunion, is a condition where the big toe deviates toward the other toes, often causing pain, difficulty with footwear, and decreased quality of life. Surgery can correct the alignment of the big toe, but during recovery the toes must be supported in the correct position so that the improvement is maintained. After this surgery, a spacer is usually placed between the big toe and the second toe for several weeks while the soft tissues heal.

Standard spacers made of folded gauze are not custom-shaped to each patient's foot, which may lead to discomfort, skin irritation, or misalignment of the other toes. To address these limitations, a new custom-made spacer has been developed using 3D printing technology. This spacer is individually designed to match each patient's foot shape, with the goal of improving comfort and maintaining proper toe alignment throughout the healing phase.

This clinical study will evaluate whether the custom-made 3D-printed spacer is better tolerated by patients than the traditional folded-gauze spacer and whether it helps maintain the corrected position of the big toe after surgery. The study will include 40 adults undergoing bunion surgery. Participants will be randomly assigned, like drawing lots, to receive either the 3D-printed spacer or the standard gauze spacer. Both spacers are applied externally during surgery and are worn continuously for five weeks as part of routine postoperative care.

Participants will attend follow-up visits at 1 week, 3 weeks, and 5 weeks after surgery. At each visit, comfort, pain, and any skin irritation caused by the spacer will be evaluated. At the final visit, toe alignment will be assessed using routine weight-bearing X-rays and clinical examination. No additional medical procedures or radiation will be required beyond standard care.

The hypothesis of this study is that the custom 3D-printed spacer will be well tolerated and will help maintain better toe alignment compared with the standard folded-gauze spacer. If successful, this personalized approach may improve recovery and patient satisfaction after bunion surgery.

DETAILED DESCRIPTION:
Hallux valgus is a common forefoot deformity characterized by lateral deviation of the hallux and medial deviation of the first metatarsal. Surgical correction is performed to restore alignment and relieve symptoms, but postoperative soft tissue healing requires mechanical support to maintain the correction during early recovery. A toe spacer is routinely used for this purpose, generally applied between the hallux and second toe for several weeks after surgery.

Traditional spacers, typically fabricated from folded gauze, are non-custom solutions that may not conform to the patient's individual anatomy. As a result, they may cause discomfort, pressure areas, or misalignment of the lesser toes. To overcome these limitations, a custom-made spacer has been designed using 3D-printing technology. The device is manufactured from thermoplastic polyurethane (TPU), a biocompatible material commonly used in orthotic applications. It is externally applied and does not enter the surgical wound. The device is intended to improve comfort and maintain postoperative hallux alignment more effectively than standard spacers.

This study is a single-center randomized controlled trial evaluating the feasibility, tolerance, and early alignment outcomes associated with the use of the custom-made 3D-printed spacer compared to standard folded-gauze spacers. Forty adult participants undergoing hallux valgus surgical correction will be randomly allocated in a 1:1 ratio to the intervention or control group through sealed opaque envelopes prepared prior to study initiation. Both interventions are non-invasive and part of routine postoperative care.

The spacer will be applied immediately after surgery and continuously maintained for five weeks. Standardized follow-up evaluations will be performed at 1, 3, and 5 weeks after surgery. Tolerance of the device will be assessed using patient-reported comfort and pain scores and clinical evaluation of skin condition, including the presence of irritation, redness, pressure marks, or ulceration. Alignment outcomes will be assessed at the final follow-up visit using routine weight-bearing radiographs and clinical examination.

The primary aim of this investigation is to assess the tolerance of the custom-made 3D-printed postoperative spacer. Secondary aims include the evaluation of hallux and lesser-toe alignment at five weeks and the documentation of spacer-related adverse events. Because this is an early clinical assessment of a new supportive postoperative device, the study is designed as a minimal-risk feasibility trial with a pragmatic sample size.

All surgical procedures and postoperative care will be conducted by fellowship-trained foot and ankle surgeons using standardized techniques. To minimize bias, allocation concealment is ensured by the envelope randomization method, follow-up timing is standardized, and imaging evaluation will be performed based on prespecified measurement criteria.

No additional imaging, radiation exposure, or medical procedures are required beyond standard postoperative care, and participation does not alter the surgical treatment plan. The study is classified under Risk Category A according to the Swiss Human Research Ordinance (HRO), as the device does not pose significant additional risks or burdens beyond normal clinical practice.

The findings of this study will provide preliminary evidence on the clinical feasibility and patient acceptance of customized postoperative spacers following hallux valgus surgery. Positive results may support future larger-scale trials designed to assess long-term clinical outcomes and validate the benefits of individualized postoperative support in forefoot surgical care.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Diagnosis of hallux valgus requiring surgical correction
* Undergoing a standard hallux valgus procedure at the study center
* Able to comply with study procedures and follow-up visits
* Signed informed consent obtained before participation

Exclusion Criteria:

* Inability to provide informed consent
* Inability to comply with study procedures or follow-up visits
* Insufficient language comprehension for study instructions
* Bilateral hallux valgus surgery planned
* Known allergy or hypersensitivity to thermoplastic polyurethane (TPU)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-04-15 (Estimated)

PRIMARY OUTCOMES:
Patient tolerance to postoperative toe spacer | 1 week, 3 weeks, and 5 weeks after surgery
  Patient tolerance measured using patient-reported comfort and pain on a 5-point Likert scale (Likert-type scale; minimum = 1, maximum = 5), where higher scores indicate better comfort and lower pain. Clinical evaluation will also assess the presence of skin irritation, redness, pressure marks or ulceration at 1 week, 3 weeks and 5 weeks after surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Assal de médecin et chirurgie du pied, Geneva, Canton of Geneva, Switzerland

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because this is a small, single-center study involving identifiable clinical and imaging data that cannot be fully anonymized while maintaining scientific value. Only aggregated results will be published in peer-reviewed journals.

REFERENCES:
- [Background] Pentikainen I, Piippo J, Ohtonen P, Junila J, Leppilahti J. Role of Fixation and Postoperative Regimens in the Long-Term Outcomes of Distal Chevron Osteotomy: A Randomized Controlled Two-by-Two Factorial Trial of 100 Patients. J Foot Ankle Surg. 2015 May-Jun;54(3):356-60. doi: 10.1053/j.jfas.2014.08.001. Epub 2014 Oct 24. PMID 25441855
- [Background] Choo YJ, Kim JH, Chang MC. Three-dimensional printing technology applied to the production of prosthesis: A systemic narrative review. Prosthet Orthot Int. 2024 Jun 18;49(3):344-352. doi: 10.1097/PXR.0000000000000366. PMID 38896537
- [Background] Saragas NP. Clinical tip: postoperative dressing for hallux valgus surgery. Foot Ankle Int. 2005 Oct;26(10):899-900. doi: 10.1177/107110070502601018. No abstract available. PMID 16221466
- [Background] Hester WA 3rd, Pedowitz DI. Postoperative Considerations in the Management of Hallux Valgus. Foot Ankle Clin. 2020 Mar;25(1):141-150. doi: 10.1016/j.fcl.2019.11.002. PMID 31997741
- [Background] Nix S, Smith M, Vicenzino B. Prevalence of hallux valgus in the general population: a systematic review and meta-analysis. J Foot Ankle Res. 2010 Sep 27;3:21. doi: 10.1186/1757-1146-3-21. PMID 20868524

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-10-15): https://cdn.clinicaltrials.gov/large-docs/56/NCT07267156/Prot_SAP_001.pdf